CLINICAL TRIAL: NCT07202117
Title: Comparing Outcomes of Collagen Biostimulatory Agents: A Randomized, Patient and Evaluator-blinded Clinical Trial Evaluating Poly-L-lactic Acid and Calcium Hydroxyapatite for Rejuvenation of the Face and Body
Brief Title: PLLA and CaHA-R for Aesthetic Rejuvenation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GAL-2025-PLLA-68
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Aesthetic
Keywords: Poly-L-Lactic-Acid; Calcium Hydroxyapatite; Injectable; Biostimulator; Aging

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Parallel-Group Clinical Trial with Unequal Allocation (2:1 ratio)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (PLLA - Sculptra® Aesthetic) (Experimental): Thirty (30) participants will receive up to three treatment of PLLA - Sculptra® Aesthetic in their face and décolleté region
  Interventions: Device: Sculptra Aesthetic
- Group B (CaHA-R - RadiesseTM) (Experimental): Fifteen (15) participants will receive up to three treatment of CaHA-R, Radiesse in their face and décolleté region
  Interventions: Device: Radiesse

INTERVENTIONS:
Device: Sculptra Aesthetic — Sculptra® Aesthetic is manufactured by Galderma Laboratories. It is a sterile, lyophilized preparation of PLLA that is biocompatible and biodegradable. Each vial contains 367.5 mg of freeze-dried powder, including 150 mg of PLLA. Prior to injection, it will be reconstituted with sterile water for injection (SWFI) and lidocaine hydrochloride (2%).
  For this study, commercial products will be used. The study products are for single use only.
  Arms: Group A (PLLA - Sculptra® Aesthetic)
Device: Radiesse — Radiesse® is manufactured by Merz Aesthetics. It is a sterile, non-pyrogenic, semi-solid injectable implant composed of synthetic CaHA suspended in a gel carrier of sterile water, glycerin, and sodium carboxymethylcellulose. Each pre-filled syringe contains 1.5 mL of product. The product includes 0.3% lidocaine for pain reduction during injection.
  For this study, commercial products will be used. The study products are for single use only.
  Arms: Group B (CaHA-R - RadiesseTM)

SUMMARY:
Skin ageing is intricately linked to collagen degradation caused by internal and external factors. External factors contributing to ageing include ultraviolet rays, smoking, heat, and air pollution, and follow a distribution across the body according to the level of exposure. Whereas internal ageing occurs as a natural consequence of physiological changes over time. As we age, both natural internal and external factors cause stress to the body. This stress damages important molecules in our skin, including proteins, fats (lipids), and DNA. One of the main proteins affected is collagen, which gives skin its strength and firmness. This loss of collagen leads to visible signs of aging such as wrinkles, thinner skin (atrophy), rough or damaged texture (elastosis), and uneven skin tone (dyschromia).

Interventions such as collagen stimulators have shown promising outcomes in stimulating cells to produce collagen, thereby improving skin elasticity and firmness. Poly-L-Lactic Acid is a biodegradable long-chain polymer of repeating units of lactic acid derived from alpha-hydroxy acid. Injecting PLLA into the deep dermis or subcutaneous tissue, stimulates collagen production through an inflammatory response, resulting in skin rejuvenation that can last between two to three years. In contrast, CaHA-R drives the regeneration of collagens, elastin, and proteoglycans with minimal immune cell recruitment and immediate volume improvement lasting around 12-18 months. To date, there have been no randomized-controlled-trials comparing the efficacy of PLLA vs CaHa-R for skin rejuvenation in the face and body.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written participant information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Participant with mild to severe skin irregularities in the bilateral cheeks and the décolletage region at baseline as assessed by both the Blinded Evaluator and Investigator (scores may differ) using the Galderma Decolletage Scale (GDS) and the Facial Laxity Rating (FLR) scale
3. Immune-competent adult pre-menopausal women 21 years of age and older.
4. Has intent to undergo treatment to improve appearance of the cheeks and décolletage.
5. Could benefit from injectable treatment to improve appearance of the cheeks and the décolletage, in the opinion of the Treating Investigator.
6. If the participant is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at Baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/ cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative UPT for women of childbearing potential at the Baseline visit.
8. Participant agrees to use the same topical cosmetic products (e.g., cleansers, moisturizers, SPF) throughout the duration of the trial, and at least for 30 days prior to enrolment.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any of the Sculptra constituents.
2. Hypersensitivity to RADIESSE, or CaHA-R-based fillers.
3. Known/previous allergy or hypersensitivity to lidocaine and other local anesthetics, e.g. amide-type anesthetics, or topical anesthetics or nerve blocking agents.
4. Previous or present severe or multiple allergies, such as anaphylaxis or angioedema, or family history of these conditions.
5. Previous surgery in or near the treatment area, including but not limited to liposuction.
6. Previous treatment/procedure in or near the treatment area:

   1. Previous permanent implant, lifting threads in the treatment area, regardless of time.
   2. Previous semi-permanent implants exemplified by CaHA-R, PLLA in treatment area, within the last 18 months of screening.
   3. Previous hyaluronic acid (HA) filler or collagen filler in the treatment area within 12 months of screening.
   4. Previous energy-based aesthetic procedures (e.g. laser, intense pulsed light, radiofrequency, HIFEM and endermologie) in the treatment area within 6 months of screening.
   5. Previous mechanical (e.g. dermabrasion, needling) or chemical aesthetic procedures (e.g. medical chemical peel) in the treatment area within 6 months of screening.
   6. Previous treatment with cryolipolysis, lipolytic treatments, ultrasound treatment, carboxytherapy or liporeduction massage in the treatment area within 6 months of screening.
   7. Previous collagenase clostridium histolyticumaaes treatment within 6 months of screening OR is planning to undergo any of these procedures affecting the treatment area, at any time during the study.
7. History of cancer or previous radiation near or on the area to be treated.
8. Heavy smokers, classified as smoking more than 12 cigarettes per day.
9. Presence of any active disease or lesions near or on the area to be treated, e.g.

   1. Inflammation, active or chronic infection in or near the treatment area
   2. Psoriasis, eczema, herpes zoster and acanthosis
   3. Cancer or precancerous condition (e.g. actinic keratosis)
   4. Severe skin laxity, flaccidity, or sagging
   5. Advanced photoaged/ photodamaged skin (e.g., advanced skin elastosis, multiple lentigo solaris lesions) or skin condition (e.g., very crinkled, very thin, fragile skin or severe skin atrophy) in the treatment area that in the Investigator's opinion could interfere with the safety or effectiveness of the study product or injection procedure.
10. Evidence of scar-related disease or delayed healing activity within 1 year prior to the baseline visit, or participants susceptible to keloid formation, or hypertrophic scarring from injectable procedures.
11. Skin coloring/bleaching/tattoo in the treatment area, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
12. Intends to initiate a weight loss program during the study (e.g., restrictive diets, GLP-1 agonists).
13. An underlying known disease, a surgical or medical condition that would expose the participant to undue risk, e.g. history of bleeding disorders, active hepatitis, active autoimmune disease such as connective tissue diseases, systemic lupus erythematosus, polymyositis, dermatomyositis, multiple sclerosis or scleroderma.
14. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., warfarin, clopidogrel, aspirin, baby aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs)), Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.
15. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (inhaled or ophthalmic corticosteroids are allowed).
16. Use of hormonal replacement therapy (HRT) unless the participant has been on a stable dose for at least 3 months prior to screening and does not plan to make any changes to the HRT regimen during the study period.
17. Use of topical corticosteroids, topical prescription retinoids in the treatment area within 1 month of the Baseline visit or systemic retinoid treatment within 6 months of the baseline visit, or plan to receive such treatment.
18. Pregnancy (confirmed by positive urine pregnancy test (UPT)/ serum pregnancy test), breast feeding or intends to become pregnant over the duration of the study.
19. Presence of any condition or situation, which in the opinion of the Treating Investigator makes the Participant unable to complete the study per protocol, e.g.

    * Participant is not likely to avoid other prohibited aesthetic treatments;
    * Participant is not likely to complete the study because of other commitments;
    * Participant is anticipated to be unavailable for visits, incapable of understanding the investigational assessments or having unrealistic expectations of treatment result;
    * Participant who has a concomitant condition (e.g., acute viral or bacterial infection with fever) that might confuse or confound study treatments or assessments.
20. Participation in any interventional clinical study within 30 days of screening.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Elasticity Measured by Cutometer | Baseline (Visit 1) to Week 40 (Visit 6)
  Change in skin elasticity parameters (net elasticity, gross elasticity, distensibility, and maximum recovery) will be measured using the Cutometer Dual MPA 580 on the cheek and décolleté.

SECONDARY OUTCOMES:
Participant Satisfaction with Treatment | Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Participant satisfaction will be assessed using a 7-point Likert scale questionnaire rating satisfaction with skin appearance after treatment (from "Very Dissatisfied" to "Very Satisfied"). Scores will be compared between groups.
Global Aesthetic Improvement Scale (GAIS) as Assessed by a Blinded Evaluator | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), Week 40 (Visit 6)
  Blinded evaluators will assess aesthetic improvement using the GAIS. The percentage of participants rated as at least "Improved" ("Improved", "Much Improved", or "Very Much Improved") compared to Baseline will be compared between groups

OTHER OUTCOMES:
Change in Facial Laxity Rating (FLR) and Galderma Decolletage Scale (GDS) as assessed by a blinded evaluator | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Facial and décolleté laxity will be rated using the 10-class Facial Laxity Rating (FLR) scale and the 5-point Galderma Decolletage Scale (GDS), assessed by a blinded evaluator.
Volume of Product Used | Baseline to Week 40 (Visit 6)
  Total volume of PLLA or CaHA-R used for each participant will be recorded to assess correlation with clinical outcomes and biophysical skin parameter changes.
Change in Skin Hydration Using the Corneometer CM 825 probe | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Changes in hydration will be measured using the Corneometer CM 825 probe on the cheek and décolleté regions at baseline and at all visits following treatments, comparison may be made between groups
Change in Transepidermal Water Loss (TEWL) Using the Tewameter TM 2 | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Changes in TEWL will be measured using the Tewameter TM 210 to evaluate barrier function improvement, comparison may be made between groups
Surface Evaluation of Living Skin Cells (SELS) using the VisioScan VC 98 | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Change in SELS will be analyzed via VisioScan VC 98 to measure skin roughness, smoothness, scaliness, desquamation, pore size, and wrinkle patterns, comparisons may be made between groups
Change in Skin Thickness as Visualized by High Frequency Ultrasonography | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Changes in skin thickness (dermis and hypodermis) will be measured using ultra-high-frequency ultrasound (Clarius L20) to quantify biostimulatory effects of each treatment, comparison may be made between groups.
3D Volumetric Analysis | Baseline to Week 40
  Volumetric changes will be measured using 3D imaging (Canfield Scientific) to assess lifting and contouring effects. Correlation with product volume will be evaluated if applicable. Comparison between volume of product used may be compared between products
Lifting Capacity via Directional Vector Analysis | Baseline to Week 40
  Lift will be assessed using vector shift analysis on 3D images. Correlation with volume used will be explored. Comparison between volume of product and lift may be compared between products
Change in Tissue Laxity Using Pinch and Slide Tests | Baseline, Week 20 (Visit 4), Week 30 (Visit 5), and Week 40 (Visit 6)
  Quantitative changes in skin laxity will be measured using digital calipers (MENTOR® MemoryGel™ Xtra).
Safety Composite Outcome | Baseline to Week 40
  Safety will be assessed based on:
  Participant-reported adverse events (via take-home diaries) Physician-reported adverse events (at all study visits) Incidence, severity, and relation to treatment will be documented and compared between groups.
Histological Evaluation of Biopsy Samples (subgroup analysis) | Baseline, Week 20 (Visit 4), and Week 40 (Visit 6)
  In consenting participants (n ≥ 15), bilateral retro-auricular biopsies will be analyzed with various stains (Masson's Trichrome, Picrosirius Red, etc.) for:
  Neocollagenesis, neovascularization, and neoelastinogenesis Dermal thickness Inflammatory response, fibrosis, or foreign body reaction Presence of procollagen, fibroblasts, eosinophils, proteoglycans, glycoproteins, hyaluronic acid
  Analysis may include comparison between products following administration of all three treatments

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No